CLINICAL TRIAL: NCT03882450
Title: Universal Screening for Vocal Fold Motion Impairment in Children Undergoing Congenital Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nikhila Raol, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00093935
Record Dates: First submitted 2019-03-08; First posted 2019-03-20 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Vocal Fold Palsy; Dysphagia; Congenital Heart Disease in Children
MeSH Terms: conditions — Vocal Cord Paralysis; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neonates with congenital cardiac disease (retrospective) (No Intervention): Medical records of all children 18 and under who underwent CCS (as defined by ICD-9-CM congenital heart disease procedure codes) from January 1, 2011 to December 31, 2016 will be reviewed. Those who developed VFMI following CCS as diagnosed on flexible fiberoptic laryngoscopy will be identified. Inpatient, outpatient and emergency department (ED) records will be studied for details on postoperative length of stay, time to diagnosis of VFMI, time to initiation of oral feeding, ED visits and readmissions for feeding/weight gain or respiratory issues, and otolaryngology intervention.
- Neonates with congenital cardiac disease (prospective) (Active Comparator): Eligible children with known congenital cardiac disease necessitating cardiothoracic surgery will undergo universal screening, i.e., laryngeal ultrasonography and flexible fiberoptic laryngoscopy with examination and video documentation of laryngeal function preoperatively (if they are not intubated and are stable enough to do so) and postoperatively with a 2.4mm flexible laryngoscope and portable ultrasound system while awake.
  Interventions: Procedure: Flexible fiberoptic laryngoscopy; Procedure: Laryngeal ultrasonography

INTERVENTIONS:
Procedure: Flexible fiberoptic laryngoscopy — Flexible fiberoptic laryngoscopy with examination and video documentation of laryngeal function preoperatively (if the participant is not intubated and is stable enough to do so) and postoperatively with a 2.4mm flexible laryngoscope will be performed.
  Arms: Neonates with congenital cardiac disease (prospective)
Procedure: Laryngeal ultrasonography — Laryngeal ultrasonography will be performed using a portable ultrasound system while the participants are awake.
  Arms: Neonates with congenital cardiac disease (prospective)

SUMMARY:
The purpose of this study is to determine how often heart or chest surgery in children leads to problems with the movement of the vocal folds.

DETAILED DESCRIPTION:
Pediatric vocal fold motion impairment (VFMI) is a well-known cause of dysphonia and dysphagia. Previous studies have demonstrated the most common etiology for pediatric VFMI is cardiothoracic surgery which is possibly due to a variety of mechanisms.The investigators hypothesize that universal screening of neonates for VMFI following congenital cardiac surgery (CCS) will lead to a more accurate incidence and earlier diagnosis of VFMI. They believe that earlier identification will lead to changes in feeding regimens that may decrease length of stay (LOS), decrease time to oral feeding, earlier otolaryngologic intervention if indicated, and decreased rates of readmission for pulmonary or feeding complications. The investigators will also use this information to design a refined algorithm for targeted screening of patients who are more likely to have VFMI based on patient and surgery characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Children 18 and younger with congenital cardiac disease necessitating surgery
* Children 18 and younger whose parents have given and signed an informed consent and HIPAA Authorization as well as the assent of the patient

Exclusion Criteria:

* History of prior cardiac surgery
* Known history of VFMI prior to evaluation
* Children 18 and younger who do not survive the immediate postoperative course will be excluded.
* Further exclusion may be determined at the discretion of the Principal Investigator.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 94 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Postoperative length of stay (retrospective) | Baseline
  The number of days of postoperative stay in the hospital will be compiled by reviewing the medical records of all children 18 and under who underwent CCS (as defined by ICD-9-CM congenital heart disease procedure codes) from January 1, 2011 to December 31, 2016.
Number of readmissions related to feeding difficulty (retrospective) | Baseline
  The number of readmissions to the hospital for feeding difficulties will be compiled by reviewing the medical records of all children 18 and under who underwent CCS (as defined by ICD-9-CM congenital heart disease procedure codes) from January 1, 2011 to December 31, 2016.
Number of readmissions related to aspiration (retrospective) | Baseline
  The number of readmissions to the hospital for aspiration will be compiled by reviewing the medical records of all children 18 and under who underwent CCS (as defined by ICD-9-CM congenital heart disease procedure codes) from January 1, 2011 to December 31, 2016.
Time to initiation of feeding therapy (retrospective) | Baseline
  The average time (in days) to start feeding therapy will be compiled by reviewing the medical records of all children 18 and under who underwent CCS (as defined by ICD-9-CM congenital heart disease procedure codes) from January 1, 2011 to December 31, 2016.
Number of participants with vocal fold motion impairment (prospective) | Baseline
  The number of study participants diagnosed with VFMI following CCS universal screening will be recorded.
Postoperative length of stay (prospective) | Up to 180 days
  The number of days of postoperative stay at the hospital will be recorded.
Time to initiation of feeding therapy (prospective) | Day 7
  The number of days to start feeding therapy will be recorded.
Number of readmissions related to aspiration (prospective) | 3 months, 6 months, 12 months
  The number of readmissions to the hospital for aspiration will be recorded.
Number of readmissions related to feeding difficulty (prospective) | 3 months, 6 months, 12 months
  The number of readmissions to the hospital for feeding difficulties will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhila Raol, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States